CLINICAL TRIAL: NCT05062850
Title: Association and Prevalence Between Geriatric Syndrome and Chronic Diseases in Nonagenarians: a Single-center Observation
Brief Title: Between Geriatric Syndrome and Chronic Disease Association and Prevalence Among Nonagenarians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Betul Gulsum Yavuz Veizi, MD, Gulhane Training and Research Hospital
Other Study IDs: 19-436
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: The Study Addressed the Most Common Geriatric Syndromes and Chronic Diseases at Age 90 Years and Older and Their Association
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — Our study does not involve an intervention. Chronic diseases and geriatric syndromes of the participants will be studied.

SUMMARY:
OBJECTİVE The world population is getting older. The most common condition in the aging population is comorbidity, which is a combination of more than one chronic disease or condition. Contrary to the traditional view that specific symptoms are characteristic of a single disease, the coexistence of multiple diseases and other age-related conditions in elderly individuals leads to what is defined as geriatric syndromes. Geriatric syndromes are quite common in the elderly population and are associated with poor quality of life, adverse health status, and increased cost. Physicians who more frequently care and manage patients with comorbid diseases and geriatric syndrome can cope better with these conditions when faced with them. It is known that the frequency of comorbidity and geriatric syndrome increases especially in the elderly. However, in the oldest age group, which is showing the fastest increase in population, these rates are not clearly known. The aim of this study is to shed light on the management of elderly patients by identifying geriatric syndromes and comorbidity prevalence, as well as chronic diseases and common geriatric syndromes, in patients 90 years of age and older who applied to the geriatric outpatient clinic.

METHOD Data of patients 90 years and older who applied to the geriatric outpatient clinic between November 2016 and January 2020 were retrospectively analyzed. The drugs used by the patients with their demographic characteristics such as age, gender, chronic diseases and geriatric syndromes were gathered. The drugs used were also obtained from the hospital-registered files and through the E-Pulse health system. Diabetes mellitus (DM), hypertension (HT), cardiovascular diseases (CVD), cerebrovascular occlusion (CVO), chronic obstructive pulmonary disease (COPD), chronic kidney disease (CKD) were recorded as chronic diseases. Mild cognitive impairment (MCI), dementia, delirium, depression, fall, incontinence, malnutrition, sleep disorders, polypharmacy, and fall were recorded as geriatric syndrome. The modified Charlson comorbidity index was used to calculate the comorbidity index.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling individuals aged 90 and over

Exclusion Criteria:

* Patients with missing data were excluded from the study

Ages: 90 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The world population is getting older. The most common condition in the aging population is comorbidity, which is the combination of more than one chronic disease or condition. In individuals 90 years of age and older, the severity of this condition is not well understood.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
prevalence | five years
  number of geriatric syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No